CLINICAL TRIAL: NCT05486312
Title: A Multi-center, Exploratory, Single-Arm, 7-week Study to Evaluate the Feasibility and Acceptability of Treatment With CT-155 in People With Schizophrenia
Brief Title: 7-week Study With CT-155 in People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CT-155-C-002
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia
Keywords: Prescription digital therapeutic (PDT); Software-as-a Medical Device (SaMD); Smartphone app; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: This is a multi-center, exploratory, single-arm study to evaluate the overall effects of use of an abbreviated version of CT-155 in adults diagnosed with schizophrenia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single arm (Experimental): Single arm acceptability and feasibility of CT-155.
  Interventions: Device: CT-155 smartphone app

INTERVENTIONS:
Device: CT-155 smartphone app — The CT-155 study app is designed to provide treatment monitoring and educational components of a full treatment cycle with CT-155. This design allows inferences to be made about the usability and acceptability of CT-155. Eligible participants will be enrolled during an in-person clinic visit on Day 1. Participants will then be directed to access the study app and perform tasks each day for the 49-day engagement period.

SUMMARY:
CT-155 is a novel prescription digital therapeutic (PDT) to treat schizophrenia

DETAILED DESCRIPTION:
CT-155 is a novel prescription digital therapeutic (PDT) being developed by Click Therapeutics, Inc. (Click) and Boehringer Ingelheim (BI) using an interactive, software-based intervention to treat schizophrenia.

This is a multi-center, exploratory, single-arm study to evaluate the feasibility and acceptability of treatment with an abbreviated version of CT-155 in adults diagnosed with schizophrenia. Eligible participants must have a diagnosis of schizophrenia per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).

Participants that meet eligibility criteria will be enrolled in the study on Day 1. The study consists of an up to 7-day screening period, a 49-day engagement period, and an up to 7-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Has outpatient treatment status of schizophrenia.
2. Is on a stable dose of antipsychotic medication(s)
3. Is the solo user of an iPhone with iPhone operating system (iOS)13 or greater capabilities or a smart phone with an Android operating system (OS) 9 or greater capabilities.
4. Is the owner of, and has regular access to, an email address.
5. Has regular access to the internet via cellular data plan and/or wifi.
6. Willing and able to receive SMS text messages on their smartphone and email messages, and understand how to use the downloaded Study App.
7. Has stable housing and has remained at the same residence for at least 12 weeks prior to screening, with no anticipated housing changes during the duration of the study

Exclusion Criteria:

1. Is currently treated with more than two antipsychotic medications.
2. Is currently treated with clozapine or haloperidol.
3. Has active prominent positive symptoms to preclude effective engagement in treatment for negative symptoms.
4. Is currently receiving or has received psychotherapy within 12 weeks prior to screening.
5. Meets either the International Classification of Diseases (ICD-10) or DSM-5 criteria for diagnoses not under investigation.
6. Has post-traumatic stress disorder (PTSD), bipolar disorder, major depressive disorder, developmental disorders, or any prominent disorder.
7. Has substance or alcohol use disorder.
8. Currently needs or will likely require prohibited concomitant medications.
9. Is currently participating in another clinical study.
10. Prior participation in the CT-155-C-001 clinical study.
11. Has suicidal ideation or behavior.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability with the study app as measured by Mobile App Rating Scale (MARS) at week 7 | MARS scale on Week 7 at the end of the treatment period
  Participants ratings of Study App quality and satisfaction as measured by the Mobile App Rating Scale (MARS) at Week 7
  The MARS is a validated 23-items rated on a 5-point anchored scale 1 being the lowest and 5 the highest

SECONDARY OUTCOMES:
Change in strength of digital working alliance from Week 3 to Week 7 as assessed by the Mobile Agnew Relationships Measure (mARM) | Change from Week 3 to Week 7 of the Mobile Agnew Relationships Measure
  To explore the establishment of a digital working alliance as assessed by the change from Week 3 to Week 7 of the Mobile Agnew Relationships Measure. The Mobile Agnew Relationships Measures is on a 7-item scale that ranges from "Strongly Disagree" as scale 1 to "Strongly Agree" as scale 7.

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Lakhan, MDPhD, FAAN, Study Chair — Click Therapeutics
Locations (10):
- United States (10):
  - CT-155 Study Center, Culver City, California
  - CT-155 Study Center, Garden Grove, California
  - CT-155 Study Center, La Habra, California
  - CT-155 Study Center, San Bernardino, California
  - CT-155 Study Center, Santa Ana, California
  - CT-155 Study Center, Chicago, Illinois
  - CT-155 Study Center, New York, New York
  - CT-155 study Center, Staten Island, New York
  - CT-155 Study Center, Beachwood, Ohio
  - CT-155 Study Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Snipes C, Dorner-Ciossek C, Hare BD, Besedina O, Campellone T, Petrova M, Lakhan SE, Pratap A. Establishment and Maintenance of a Digital Therapeutic Alliance in People Living With Negative Symptoms of Schizophrenia: Two Exploratory Single-Arm Studies. JMIR Ment Health. 2025 Jan 27;12:e64959. doi: 10.2196/64959. PMID 39869902